CLINICAL TRIAL: NCT02949895
Title: A Phase 1 Study of the Safety and Tolerability of BMS-986012 in Subjects With Small Cell Lung Cancer
Brief Title: Study of BMS-986012 in Subjects With Small Cell Lung Caner
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA001-045
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Escalation Dose 1 (Experimental): BMS-986012 Dose Escalation Dose 1
  Interventions: Drug: BMS-986012
- Dose Escalation Dose 2 (Experimental): BMS-986012 Dose Escalation Dose 2
  Interventions: Drug: BMS-986012
- Chemotherapy Combination (Experimental): BMS-986012 + Cisplatin + Etoposide
  Interventions: Drug: BMS-986012; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: BMS-986012
Drug: Cisplatin
  Arms: Chemotherapy Combination
Drug: Etoposide
  Arms: Chemotherapy Combination

SUMMARY:
A study to evaluate safety and tolerability of BMS-986012 in patients with small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

* Histological or cytological confirmed small cell lung cancer (SCLC)
* Eastern Cooperative Oncology Group Performance Status 0-1
* at least one measurable lesion that is not amenable to resection.
* Adequate organ function

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases
* Grade ≥ 2 peripheral neuropathy
* Uncontrolled or significant cardiac disease
* Active or chronic infection with Human Immunodeficiency Virus(HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV)

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 2 years
Number of participants with serious adverse events (SAEs ) | Up to 2 years
Number of Discontinuations due to AEs | Up to 2 years
Number of Deaths due to AEs | Up to 2 years
Number of participants with laboratory toxicity grade shift from baseline | Up to 2 years

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Time of maximum observed serum concentration(Tmax) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration(AUC(0-T)) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Observed serum concentration at the end of a dosing interval(Ctau) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Area under the concentration-time curve in 1 dosing interval(AUC(TAU)) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Characterization of Immunogenicity as measured by Anti-Drug Antibodies (ADA) | Cycle 1(each cycle is 21 days) Day 1 up to 60 days after last dose
Best overall response (BOR) | Cycle 1(each cycle is 21 days) Day 1 up to approximately 2 years
Duration of response (DOR) | Cycle 1(each cycle is 21 days) Day 1 up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Takatsuki-shi, Osaka
  - Local Institution, Chuo-ku, Tokyo

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx